CLINICAL TRIAL: NCT04063839
Title: Management of Hepatitis C Virus Infection Among People Who Inject Drugs in a Low-threshold Setting: Efficacy of Direct-acting Antiviral Treatment and the Risk of Reinfection
Brief Title: HCV Treatment in a Low-threshold Clinic
Acronym: Prindsen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Olav Dalgard, Professor, University Hospital, Akershus
Other Study IDs: 17_120
Record Dates: First submitted 2019-06-27; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hepatitis C; Substance Use Disorders
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders | interventions — elbasvir-grazoprevir drug combination; Sofosbuvir; ledipasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma collected at baseline and stored frozen -70 C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Elbasvir / Grazoprevir Oral Tablet — HCV treatment according to Norwegian guidelines
  Other Names: sofosbuvir; ledipasvir

SUMMARY:
This is a cohort of people who inject drugs with chronic HCV infection. Patients are seen at a low-threshold clinic. All patients are offered treatment for HCV and subsequently followed for to years

DETAILED DESCRIPTION:
This is a cohort of people who inject drugs with chronic HCV infection. Patients are seen at a low-threshold clinic. All patients are offered treatment for HCV and subsequently followed for to years

Inclusion Consenting patients older than 18 years attending the low threshold HCV clinic in Oslo

The primary aims are to assess the efficacy (SVR rate) of DAA treatment among PWID treated in a low-threshold primary care setting (Work Package 1) and to estimate the incidence HCV reinfection f

The secondary aims are to:

* Evaluate adherence to DAA treatment (Work Package 1)
* Identify factors associated with SVR and adherence (Work Package 1)
* Characterize reinfection using next generation sequencing (Work Package 2)
* Identify factors associated with reinfection (Work Package 2)
* Evaluate changes in recent injecting risk behaviours longitudinally (Work Package 2)
* Identify factors associated with changes in risk behaviours (Work Package 2)

The hypothesis is that high SVR rates and good treatment adherence will be achieved in PWID treated for HCV infection in a low-threshold primary health care setting. Further,it is anticipated that the incidence of reinfection will be 5-10/100 PY and associated with younger age, low education level and ongoing injecting risk behaviours.

The study will include 300 patients and are close to achieving that aim the summer of 2019

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive Attending the low-threshold HCV clinic in Oslo

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ever injected drugs (100%) OAT (70%) Recent injecting drug use (70%)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sustained virological response | 12 weeks
  HCV RNA undetectable 12 weeks post treatment
Reinfection | 2 years
  HCV RNA detectable after SVR 12 in a patient who injected drugs post SVR 12

CONTACTS AND LOCATIONS:
Overall Officials: Olav Dalgard, MD PhD, Study Chair — University Hospital, Akershus
Locations (1):
- AkershusUH, Lørenskog, Select A State Or Province, Norway

IPD SHARING:
Plan to Share IPD: Undecided
depends on patient privacy decission